CLINICAL TRIAL: NCT03695380
Title: A Phase Ib Study of Cobimetinib Administered in Combination With Niraparib, With or Without Atezolizumab, To Patients With Advanced Platinum-sensitive Ovarian Cancer
Brief Title: A Clinical Study of Cobimetinib Administered in Combination With Niraparib, With or Without Atezolizumab to Patients With Advanced Platinum-sensitive Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO40482; 2018-000631-27 (EudraCT Number)
Record Dates: First submitted 2018-09-30; First posted 2018-10-04 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: OVARIAN CANCER
MeSH Terms: conditions — Ovarian Neoplasms | interventions — cobimetinib; niraparib; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Cobimetinib - Niraparib (Experimental): Stage 2 - Patients will receive cobimetinib PO QD on Days 1-21 (21/7 schedule) in combination with niraparib PO QD on Days 1-28 of each 28-day cycle at the established dose for the doublet regimen in Stage 1, Cohort 1.
  Interventions: Drug: Cobimetinib; Drug: Niraparib
- Arm B: Cobimetinib - Niraparib - Atezolizumab (Experimental): Stage 2 - Patients will receive cobimetinib PO QD on Days 1-21 (21/7 schedule) in combination with niraparib QD on Days 1-28 at the established doses for the triplet regimen in Stage 1,Cohort 2 plus atezolizumab by IV infusion at the fixed dose of 840 mg on Days 1 and 15 (+/-3 days) of each 28-day cycle.
  Interventions: Drug: Cobimetinib; Drug: Niraparib; Drug: Atezolizumab
- Cohort 1 - Cobimetinib - Niraparib (Experimental): Stage 1 - Patients in Cohort 1 will be treated with cobimetinib plus niraparib.
  Cobimetinib: Patients will receive a starting dose of 60 mg by mouth (PO) daily (QD) on Days 1-21 of each 28-day cycle.
  Niraparib: Patients will receive a starting dose of 200 mg of niraparib PO QD on Days 1-28 of each 28-day cycle.
  Interventions: Drug: Cobimetinib
- Cohort 2 - Cobimetinib - Niraparib - Atezolizumab (Experimental): Stage 1 - Patients in Cohort 2 will be treated with cobimetinib plus niraparib and atezolizumab.
  Cobimetinib: Patients will receive a starting dose of 60 mg by mouth (PO) daily (QD) on Days 1-21 of each 28-day cycle.
  Niraparib: Patients will receive a starting dose of 200 mg of niraparib PO QD on Days 1-28 of each 28-day cycle.
  Atezolizumab: Patients will also receive atezolizumab administered as an IV infusion at a fixed dose of 840 mg on Days 1 and 15 (+/-3 days) of each 28-day cycle.
  Interventions: Drug: Cobimetinib

INTERVENTIONS:
Drug: Cobimetinib — Cobimetinib will be administered at a starting dose of 60 mg by mouth (PO) daily (QD) on Days 1-21 of each 28-day cycle (Stage 1) and PO QD on Days 1-21 (21/7 schedule) at the established dose for the doublet regimen in Stage 1 (Stage 2).
Drug: Niraparib — Niraparib will be administered at a starting dose of 200 mg of niraparib PO QD on Days 1-28 of each 28-day cycle (Stage 1) and PO QD on Days 1-28 of each 28-day cycle at the established dose for the doublet regimen in Stage 1 (Stage 2).
  Arms: Arm A: Cobimetinib - Niraparib; Arm B: Cobimetinib - Niraparib - Atezolizumab
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at the fixed dose of 840 mg on Days 1 and 15 (+/-3 days) of each 28-day cycle (Stages 1 and 2).
  Arms: Arm B: Cobimetinib - Niraparib - Atezolizumab

SUMMARY:
The study will include a safety run-in phase (Stage 1) and a randomization phase (Stage 2).

The purpose of Stage 1 is to evaluate the safety of cobimetinib when administered in combination with niraparib (Cohort 1) and cobimetinib with niraparib plus atezolizumab (Cohort 2).

Stage 1 will enable patient enrollment in the randomized phase of the study (Stage 2) with both regimens at the recommended dose levels from Stage 1.

Stage 2 is a randomized, dose-expansion phase, evaluating clinical outcomes in patients with advanced platinum-sensitive ovarian cancer.

All patients will continue to receive study treatment until disease progression (according to "Response Evaluation Criteria in Solid Tumors" (RECIST), Version 1.1, unacceptable toxicity, death, or patient or investigator decision to withdraw, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria

* Ability to comply with the study protocol, in the investigator's judgment
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures, including the completion of patient-reported outcome questionnaires
* Histological diagnosis of high-grade serous or Grade 2 or Grade 3 endometrioid epithelial ovarian, fallopian tube, or primary peritoneal cancer
* Previous treatment with a minimum of one and a maximum of two prior platinum based treatment regimens
* Platinum-sensitive disease
* Availability of tumor biopsy tissue prior to first dose of study treatment with confirmation by the central laboratory that the sample is not only of adequate quality but also assignable to a molecularly defined subgroup based on breast cancer susceptibility gene (BRCA) and loss of heterozygosity (LOH) status
* Measurable disease, as defined by Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1)
* Adequate hematologic and organ function
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* Resolved or stabilized toxicities resulting from previous therapy to Grade 1
* Negative HIV test at screening
* Negative hepatitis B surface antigen and total hepatitis B core antibody (HBcAb) test, or positive total HBcAb test followed by quantitative hepatitis B virus (HBV) DNA < 500 IU/mL test at screening
* Negative hepatitis C virus (HCV) antibody test, or positive HCV antibody test followed by a negative HCV RNA test at screening
* For women of childbearing potential: Women must remain abstinent or use two contraceptive methods with a failure rate of <1% per year during the treatment period and for at least 3 months after the last dose of cobimetinib, 6 months after the last dose of niraparib, and 5 months after the last dose of atezolizumab. Women must refrain from donating eggs during this same period

Exclusion Criteria

* Prior treatment with mitogen-activated protein kinase inhibitor, polyadenosine diphosphate-ribose polymerase inhibitor, or immune checkpoint inhibitor therapies
* Prior chemotherapy, hormonal therapy, radiotherapy, antibody therapy, or other immunotherapy, gene therapy, vaccine therapy, or treatment with experimental drugs within 14 days prior to first dose of study treatment
* Treatment with systemic immunostimulatory agents within 28 days or 5 half-lives of the drug prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication 14 days prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the study
* History of other malignancy that could affect compliance with the protocol or interpretation of results, or known to have potentially fatal outcome
* Symptomatic and/or untreated central nervous system metastases
* Surgical procedure, significant traumatic injury within 14 days prior to enrollment, or anticipation of need for major surgical procedure during the study
* Minor surgical procedure within 3 days
* History or evidence of retinal pathology on ophthalmic examination
* Left ventricular ejection fraction below institutional lower limit of normal
* History of clinically significant cardiovascular dysfunction
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on the screening chest computed tomography scan
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk for bleeding
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins, or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of the cobimetinib or niraparib formulation
* Active or history of autoimmune disease or immune deficiency including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, anti-phospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barre syndrome, or multiple sclerosis
* Uncontrolled serious medical or psychiatric illness
* History of malabsorption or other condition that would interfere with absorption of oral study drugs, including preexisting duodenal stent or ongoing intestinal obstruction
* Active tuberculosis
* Severe infection within 14 days prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 7 days prior to initiation of study treatment
* Treatment with a live, attenuated influenza vaccine within 28 days prior to study treatment initiation, at any time during the study, and for at least 5 months after the last dose of study drug
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Previous treatment with strong CYP3A inhibitors (such as ketoconazole and clarithromycin), strong CYP3A inducers (such as carbamazepine and phenytoin), and moderate CYP3A inducers (such as efavirenz, modafinil) within 7 days prior to the initiation of study treatment or with ongoing requirements for these medications
* Pregnancy or breastfeeding, or intention to become pregnant during the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Number of patients reporting Adverse Events (AEs) | From baseline up to 48 months
  The safety profiles of Cobimetinib plus Niraparib and Cobimetinib plus Niraparib plus Atezolizumab will be evaluated in terms of number of patients reporting serious and non-serious AEs with severity graded according to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI - CTCAE v5.0)
Change from baseline in targeted clinical laboratory test results | From baseline up to 48 months
  The safety profiles of Cobimetinib plus Niraparib and Cobimetinib plus Niraparib plus Atezolizumabwill be evaluated in terms of number of patients reporting change from baseline in targeted clinical laboratory test results.
Investigator-assessed confirmed objective response rate (ORR) | From baseline up to 48 months
  The efficacy profiles of Cobimetinib plus Niraparib and Cobimetinib plus Niraparib plus Atezolizumab will be evaluated in terms of investigator-assessed confirmed ORR, as determined using RECIST v1.1 in the Intention To Treat (ITT) population and in molecularly defined subgroups by loss of heterozygosity (LOH) status.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From Baseline up to 48 months
  The efficacy profiles of Cobimetinib plus Niraparib and Cobimetinib plus Niraparib plus Atezolizumab will be evaluated in terms of PFS after randomization, defined as the time from randomization to the first occurrence of disease progression or relapse, as determined by the investigator using RECIST v1.1, or death from any cause during the study, whichever occurs first, in the ITT population and in the molecularly defined subgroups by LOH status.
Duration of response (DOR) | From baseline up to 48 months
  The efficacy profiles of Cobimetinib plus Niraparib and Cobimetinib plus Niraparib plus Atezolizumab will be evaluated in terms of DOR, defined for patients achieving at least one confirmed Partial Response (PR), which is measured from the first observation of a Complete Response (CR) or a PR to the time of disease progression in the ITT population and in the molecularly defined subgroups by LOH status.
Overall survival (OS) | From baseline up to 48 months
  The efficacy profiles of Cobimetinib plus Niraparib and Cobimetinib plus Niraparib plus Atezolizumab will be evaluated in terms of OS after randomization, defined as the time from randomization until death from any cause in the ITT population and in the molecularly defined subgroups by LOH status.
Plasma concentration of cobimetinib and niraparib | Arm A: Day 15 of Cycle 1 and 2 - Arm B: Day 15 of Cycle 1
  The Pharmacokinetic (PK) profile of cobimetinib plus niraparib is evaluated in terms of Plasma concentration at specified timepoints.
Serum concentration of atezolizumab | Day 1 of Cycle 1, 2 and 3 and at treatment discontinuation visit, up to 48 months
  The PK profile of cobimetinib plus niraparib plus atezolizumab will be evaluated in terms of Serum concentration of atezolizumab at specified timepoints (Arm B only).
Number of patients with Anti-Drug Antibodies (ADA) | Day 1 of Cycle 1, 2 and 3 and at treatment discontinuation visit, up to 48 months
  The immunogenicity profile of Atezolizumab is evaluated in terms of number of patients with ADA at baseline and during the study.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (9):
  - University of Arizona Cancer Center, North, Tucson, Arizona
  - Moores Cancer Center at UC San Diego Health, La Jolla, California
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Florida Hospital Cancer Institute; Clinical Research Department, Orlando, Florida
  - Medical College of Georgia; Obstetrics & Gynecolog, Augusta, Georgia
  - Washington University School of Medicine; Dept of Medicine/Div of Medical Oncology, St Louis, Missouri
  - Stephenson Cancer Center Investigational Pharmacy, Oklahoma City, Oklahoma
  - Tennessee Oncology; Sarah Cannon Research Institute, Nashville, Tennessee
  - Medical College of Wisconsin; Department of Obstetrics and Gynecology, Milwaukee, Wisconsin
- Italy (3):
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Fondazione Policlinico Universitario "A. Gemelli"; Unità di Fase 1: Unità di Farmacologia Clinica, Rome, Lazio
  - Istituto Europeo di Oncologia; Svil. Nuovi Farmaci per Terapie Innovative, Milan, Lombardy
- Spain (8):
  - Centro Oncologico de Galicia COG; Medical Oncology, A Coruña, LA Coruña
  - Hospital Universitari Vall dHebron; Oncology, Barcelona
  - ICO Girona, Girona
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Clinica Universidad de Navarra Madrid; Servicio de Oncología, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Clinico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Clínico Universitario de Valencia; Servicio de Oncología, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Mutch D, Voulgari A, Chen XM, Bradley WH, Oaknin A, Perez Fidalgo JA, Montosa FG, Herraez AC, Holloway RW, Powell MA, Nowicka M, Schaefer G, Merchant M, Yan Y. Primary results and characterization of patients with exceptional outcomes in a phase 1b study combining PARP and MEK inhibition, with or without anti-PD-L1, for BRCA wild-type, platinum-sensitive, recurrent ovarian cancer. Cancer. 2024 Jun 1;130(11):1940-1951. doi: 10.1002/cncr.35222. Epub 2024 Jan 30. PMID 38288862